CLINICAL TRIAL: NCT06140394
Title: The Effect of Low-Level Laser Therapy as an Adjunct to Non-surgical Therapy on Inducible Nitrous Oxide Synthase Salivary Levels in Different Age Groups of Chronic Periodontitis Patients (A Randomized Clinical Trial)
Brief Title: The Effect of Low-Level Laser Therapy as an Adjunct to Non-surgical Therapy in Different Age Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Alaa Allah Hesham, Bachelor's Degree (research assistant), Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P-ME-23-04
Record Dates: First submitted 2023-11-12; First posted 2023-11-20 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Periodontal Inflammation
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- old age group (Active Comparator): old age group above 60 years old
  Interventions: Other: diode laser; Other: non surgical scaling
- young aged group (Placebo Comparator): young age group below 40 years old
  Interventions: Other: diode laser; Other: non surgical scaling

INTERVENTIONS:
Other: diode laser — low level diode therapy
Other: non surgical scaling — non surgical scaling using ultrasonic

SUMMARY:
the summary is to evaluate The Effect of Low-Level Laser Therapy as an Adjunct to Non-surgical Therapy on Inducible Nitrous Oxide Synthase Salivary Levels in Different Age Groups of Chronic Periodontitis Patients

DETAILED DESCRIPTION:
2 ml of unstimulated saliva will be collected using spitting method, the collected samples will then be analyzed using Elisa technique for salivary Inducible nitrous oxide synthase levels.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* aged below 40 or above 60
* periodontitis stage 2
* no tooth loss due to periodontitis

Exclusion Criteria:

* smoking habits
* history of antibiotics
* history of systemic diseases

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
clinical parameters (gingival index) | 6 months
  measurement if the gingival index using scoring system. A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation.
clinical parameters (clinical attachment loss) | 6 months
  measurement of clinical parameters clinical attachment loss in millimeters

SECONDARY OUTCOMES:
assessment of inducible nitrous oxide synthase levels | 3 months
  measurement of inducible nitrous oxide synthase levels in different age groups before the procedure and after using Elisa kit.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa H hesham mosa, bachelor's, Study Chair — Faculty of Dental Medicine for Girls; hamdy H nassar, Principal Investigator — Faculty of Dental Medicine for Girls; amal AA ali, Study Director — Faculty of Dental Medicine for Girls
Locations (2):
- Egypt (2):
  - Al-Azhar University, Cairo, Nasrcity Nasr Street
  - Hamdy Nassar, Cairo